CLINICAL TRIAL: NCT06482307
Title: Molecular Imaging of DNA Damage Response by [18F]-Olaparib PET
Acronym: [18F]-olaparib
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19310
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Head and Neck Squamous Cell Carcinoma (HNSCC)
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Intervention Model Description: patients with HNSCC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stage I (Experimental): Five patients with HNSCC will undergo a dynamic [18F]-olaparib PET during 30 min, followed by a static whole body PET scans at 120 min post-injection of [18F]-olaparib.
  Interventions: Diagnostic Test: [18F]-olaparib PET scan
- Stage II (Experimental): After determination of the most optimal time point for imaging, five patients with HNSCC scheduled for chemoradiotherapy will undergo serial [18F]-olaparib PET at baseline (i.e. prior to treatment initiation) and a second scan during the first week of chemoradiotherapy. Patients in stage II will undergo a study biopsy in the first week of chemoradiotherapy to evaluate changes in PARP protein expression.
  Interventions: Diagnostic Test: [18F]-olaparib PET scan

INTERVENTIONS:
Diagnostic Test: [18F]-olaparib PET scan — The IMP investigated is [18F]Olaparib, a radiolabelled PARP inhibitor suitable for PET imaging.

SUMMARY:
This is a single-centre, non-randomized, two-stage design, proof-of-concept study evaluating the radiolabelled PARP inhibitor [18F]-olaparib als potential tracer for imaging of tumour PARP expression by PET.

ELIGIBILITY:
Inclusion Criteria:

1. Patients >18y, with biopsy-proven HPV-negative HNSCC, or patients >40y with HPV-positive HNSCC and high-risk features (i.e. > 10 smoke packs/year AND ≥N2b)
2. Treatment with chemoradiotherapy using platinum-based chemotherapy is anticipated
3. Recent archival tumour tissue (<8 weeks prior to inclusion) should be available with suffi-cient residual material for determination of tumour PARP1 levels
4. Presence of a tumour lesion ≥10 mm in diameter
5. ECOG performance status 0-2
6. Negative pregnancy test in women with childbearing potential
7. Life expectancy >3 months
8. Signed written informed consent and able to comply with the protocol
9. For stage II only: re-biopsy should be deemed feasible by the investigators (assessed by head-and-neck surgeon)

Exclusion Criteria:

1. Recent treatment with PARP inhibitors or other investigational therapies <30 days.
2. Presence of significant co-morbidities that make participation in the study undesirable according to the treating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Dosimetry assessment | 6-12 months
  Assess dosimetry, most optimal time point for imaging (Stage I), and safety of [18F]olaparib PET (Stage I + II)
Correlation between tumour uptake and expression | 12-18 months
  Determine the correlation between tumour [18F]-olaparib uptake and tumour PARP-1 expression levels on tumour biopsy (Stage I + II).

SECONDARY OUTCOMES:
Evaluation of changes in tumour uptake | 12-18 months
  Evaluate changes in tumour [18F]-olaparib uptake, as a read-out of DNA damage, during treatment with platinum-based chemoradio-therapy, and its correlation with changes in PARP protein expression (Stage II).

CONTACTS AND LOCATIONS:
Overall Officials: Michel van Kruchten, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided